CLINICAL TRIAL: NCT00672386
Title: A 12-Week, Double-Blind, Randomized, Placebo-Controlled Study in Type 2 Diabetes Mellitus Subjects to Evaluate the Efficacy, Safety and Tolerability of MTP Inhibitor JNJ-16269110 (R256918)
Brief Title: A Study of the Safety and Effectiveness of a R256918 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013051; CR013051
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Nutritional and Metabolic Diseases
Keywords: Diabetes; Type 2 Diabetes; Adult-Onset Diabetes Mellitus; Metabolic Syndrome; HbA1c; Body Weight; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Nutritional and Metabolic Diseases; Metabolic Syndrome; Body Weight | interventions — Metformin; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 001 (Experimental): JNJ16269110 5 mg twice daily for 12 weeks
  Interventions: Drug: JNJ16269110; Drug: Metformin; Other: Dietary Counseling
- 002 (Experimental): JNJ16269110 10 mg twice daily for 12 weeks
  Interventions: Drug: JNJ16269110; Drug: Metformin; Other: Dietary Counseling
- 003 (Experimental): JNJ16269110 15 mg twice daily for 12 weeks
  Interventions: Drug: JNJ16269110; Drug: Metformin; Other: Dietary Counseling
- 004 (Placebo Comparator): Placebo twice daily for 12 weeks
  Interventions: Drug: Placebo; Drug: Metformin; Other: Dietary Counseling

INTERVENTIONS:
Drug: JNJ16269110 — 5 mg twice daily for 12 weeks
  Arms: 001
Drug: JNJ16269110 — 10 mg twice daily for 12 weeks
  Arms: 002
Drug: JNJ16269110 — 15 mg twice daily for 12 weeks
  Arms: 003
Drug: Placebo — twice daily for 12 weeks
  Arms: 004
Drug: Metformin — Participants will continue taking metformin at the same dose and according to the same dosing regimen as before the study.
Other: Dietary Counseling — Participants will receive dietary counseling at Screening, Week 4, 8, 12, and will be instructed to remain on a calorically appropriate diet with a maximum of 30% of calories derived from fat (in accordance with local practice guidelines for the treatment of type 2 diabetes mellitus) during the entire study.

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of 12 weeks of treatment with R256918 in patients with Type 2 Diabetes Mellitus who are taking metformin. The primary measure of effectiveness is the change in concentration of glycated hemoglobin (HbA1c) during treatment. Glycated hemoglobin is a substance in red blood cells that is formed when blood sugar (glucose) attaches to hemoglobin and is a measure of diabetic status. Additional measures include fasting glucose, and lipid levels, and body weight. Safety assessments performed during the trial include laboratory tests, vital sign measurements, and adverse event reporting.

DETAILED DESCRIPTION:
This is a randomized (assigned study drug by chance), double-blind (both the patient and investigator do not know whether patient is assigned to receive study drug or placebo), placebo-controlled study involving patients with Type 2 Diabetes Mellitus who are taking metformin. Patients are randomized to one of 4 treatment groups and receive study drug (R256918: 5 mg, 10 mg, or 15 mg twice daily) or placebo for a period of 12 weeks. The study consists of a screening period, a baseline visit, the treatment period of 12 weeks, and a follow-up visit. During the treatment period, patients visit the center every two weeks. On each visit, patients come to the clinic after 8 hours fasting. Effectiveness assessments from a blood sample include levels of fasting hemoglobin type A1c (HbA1c), glucose, cholesterol, triglycerides, insulin, C-peptide, and gastrointestinal hormones. Patients monitor their fasting blood glucose and record it in a diary. Insulin sensitivity and beta cell (insulin-producing cells in the pancreas) function are evaluated. Waist and hip circumference are measured. Safety evaluations, including incidence of adverse events, clinical laboratory results, vital signs, and electrocardiograms, are performed during the study. Patients complete a questionnaire related to treatment satisfaction of study medication. Patients receive dietary counseling and will be instructed to remain on a calorically appropriate diet with a maximum of 30 percent (%) of calories derived from fat (in accordance with local practice guidelines for the treatment of type 2 diabetes mellitus), during the entire study. Patients continue taking metformin in the same dose and according to the same dosing regimen as before the study. The overall duration of the study for each patient is approximately 18 weeks. The study will evaluate the effect of R25691 on glucose-dependent insulin secretion, weight loss and changes in insulin sensitivity and tolerability in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* History of Type 2 Diabetes Mellitus and treated with a stable dose of metformin for at least 2 months
* Women must be postmenopausal or surgically incapable of childbearing or if sexually active, be practicing an effective method of birth control
* BMI between 25 and 45 kg/m2
* HbA1c between 7% and 10%, inclusive
* Fasting plasma glucose not exceeding 240mg/dL (13.3mmol/L)

Exclusion Criteria:

* Diabetes other than type 2 diabetes mellitus
* Treatment with oral anti-diabetic agents (other than metformin) or insulin during the 12 weeks before baseline visit
* History of intolerance or hypersensitivity to sulfonylurea or sitagliptin
* History of clinically significant gastrointestinal, hepatic or cardiovascular disease
* Active proliferative diabetic retinopathy
* History of diabetic gastroparesis
* concurrent use of systemic corticosteroid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c from baseline to week 12 | baseline, week 4, 6, 8, 10 and 12

SECONDARY OUTCOMES:
Changes in fasting plasma glucose | every 2 weeks
Changes in body weight | every 2 weeks
Changes in plasma lipids | baseline, week 6 and 12
Changes in systolic and diastolic blood pressure | every 2 weeks
Changes in insulin sensitivity and beta cell function (homeostatic model assessment 2 - HOMA-2 and MMTT); Changes in GLP-1 (glucagon-like peptide 1) and PYY (peptide tyrosine tyrozine) levels in the MMTT; Changes in insulin and glucagon | baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (62):
- Edegem, Belgium
- Denmark (2):
  - Hellerup
  - Vipperroed
- Finland (4):
  - Helsinki
  - Hyvinkää
  - Kuopio
  - Oulu
- Germany (7):
  - Buch
  - Dresden
  - Düsseldorf
  - Hamburg
  - Mainz
  - München
  - Ulm
- India (6):
  - Bangalore
  - Chennai
  - Hyderabad
  - Mumbai
  - Nagpur
  - Pune
- Netherlands (7):
  - Breda
  - Eindhoven
  - Leiden
  - Nijmegen
  - Rotterdam
  - Velp Gld
  - Zoetermeer
- Norway (2):
  - Oslo
  - Paradis
- Poland (11):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Kutno
  - Lodz
  - Olsztyn
  - Pruszków
  - Torun
  - Warsaw
  - Wroclaw
  - Zielona Góra
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Saratov
- Sweden (7):
  - Ängelholm
  - Gothenburg
  - Härnösand
  - Linköping
  - Lund
  - Örebro
  - Stockholm
- United Kingdom (12):
  - Bangor
  - Belfast
  - Birmingham
  - Cambridge
  - Cardiff
  - Clydebank
  - Dundee
  - Liverpool
  - London
  - Randalstown
  - Reading
  - Salford